CLINICAL TRIAL: NCT00640705
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Diclofenac Sodium Patch for the Topical Treatment of Pain Due to Mild to Moderate Ankle Sprain.
Brief Title: Diclofenac Patch for Treatment of Mild to Moderate Ankle Sprain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cerimon Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Dan Levitt, MD, Cerimon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCF-002
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Topical diclofenac sodium patch
  Interventions: Drug: diclofenac sodium
- B (Placebo Comparator): Topical patch identical in appearance to active comparator, except without diclofenac sodium
  Interventions: Drug: Matching placebo patch

INTERVENTIONS:
Drug: diclofenac sodium — 15 mg (1%) topical patch; measuring 7 cm by 10 cm; applied once daily
  Other Names: diclofenac
  Arms: A
Drug: Matching placebo patch — Matching placebo patch, containing identical constituents to the active comparator except for diclofenac sodium; measuring 7 cm by 10 cm; applied once daily
  Other Names: placebo comparator
  Arms: B

SUMMARY:
The primary purpose of this study is to assess the effectiveness of once daily application of a diclofenac sodium patch to the skin near or over the painful area. In this study, the location being studied will be either the left or right ankle.

The secondary purpose of this study is to assess the safety and tolerability of a diclofenac patch on the skin.

DETAILED DESCRIPTION:
Cerimon Pharmaceuticals is investigating a topical patch formulation of diclofenac sodium containing 15 mg of diclofenac sodium for the local treatment of acute musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Has sustained a painful Grade 1 or 2 ankle sprain (Appendix H) no more than 48 hours prior to study entry
* Presence of pain of at least 5, with a maximum of 9, on an 11-point Numerical Rating Scale (NRS)

Exclusion Criteria:

* Grade 3 ankle sprain or bilateral sprain (see Appendix H)
* Previous injury to the same ankle within 3 months prior to current injury
* Aspirin or short half-life NSAID use within 12 hours, or longer half-life NSAID use within 24 hours prior to study entry (Appendix B)
* Opioid use within 24 hours prior to study entry
* Topical treatment, other than ice packs, applied to the painful region since time of injury
* A history of peptic ulcer disease within 1 year of study entry, any history of gastrointestinal bleeding or coagulation disorder
* A history of, or evidence for, underlying disease in the injured ankle, such as osteoarthritis or gout
* Clinically significant, poorly controlled pulmonary, gastrointestinal, hepatic, renal, endocrine, or cardiovascular disease
* A history of hypersensitivity to diclofenac or diclofenac-containing products
* A history of intolerance to acetaminophen (rescue medication in this trial)
* A history of skin sensitivity to adhesives (e.g. adhesive tape)
* Pregnant or breastfeeding women and women of child-bearing potential not using effective means of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of diclofenac in subjects with mild to moderate ankle sprain. | 7 days

SECONDARY OUTCOMES:
Assess the safety and tolerability of diclofenac in subjects with mild to moderate ankle sprain. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, MD, Study Director — Cerimon Pharmaceuticals
Locations (1):
- PPD, Austin, Texas, United States